CLINICAL TRIAL: NCT05683054
Title: A Non-inferiority Study on Dose Reduction of Adalimumab in Psoriasis Patients Who Are Overtreated
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDM-ADA2019
Record Dates: First submitted 2022-12-21; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: A prospective, single blinded, randomized, non-inferiority study
Who Masked: Outcomes Assessor
Masking Description: PASI and IGA score will be performed by a blinded and independent physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dosing group (Active Comparator): In the standard based arm, patients will continue to receive adalimumab according to the standard dosing schedule of 40 mg every other week (maintenance phase).
  Interventions: Procedure: Venapuncture; Other: Dermatology Life Quality Index (DLQI); Other: EQ-5D-5L questionnaire; Procedure: Dried blood spot sampling
- Dose tapering group (Active Comparator): In the dose tapering arm, adalimumab dosing frequency will be lowered to 40 mg every 3 weeks in patients who have supratherapeutic serum trough levels of adalimumab at three consecutive measurements.
  Interventions: Biological: Dose tapering of adalimumab in patients with supratheurapeutic serum trough levels; Procedure: Venapuncture; Other: Dermatology Life Quality Index (DLQI); Other: EQ-5D-5L questionnaire; Procedure: Dried blood spot sampling

INTERVENTIONS:
Biological: Dose tapering of adalimumab in patients with supratheurapeutic serum trough levels — In the dose tapering arm, adalimumab dosing frequency will be lowered to 40 mg every 3 weeks in patients who have supratherapeutic serum trough levels of adalimumab (33% reduction). If patients still have a good clinical response and supratherapeutic adalimumab serum trough levels, will be further tapered to a dose regimen of 1 subcutaneous injection (40mg) every 4 weeks (50% dose reduction).
  Arms: Dose tapering group
Procedure: Venapuncture — Blood samples will be collected to determine the serum trough levels and anti-drug antibodies of adalimumab
Other: Dermatology Life Quality Index (DLQI) — The impact of the disease on the patient will be assessed using the dermatology life quality index (DLQI).
Other: EQ-5D-5L questionnaire — The EQ-5D-5L which is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments will be assessed.
Procedure: Dried blood spot sampling — A subset of patients will sample additionally by using dried blood sampling after the first drug injection post-inclusion.

SUMMARY:
Recently, the optimal therapeutic serum trough level range of adalimumab was defined between 3,5 and 7,0 µg/ml in patients with plaque type psoriasis. An adalimumab serum through level above this therapeutic range did not add to clinical response. Based on this therapeutic window, the introduction of dose adjustments based on serum trough levels (therapeutic drug monitoring) will be further validated in a prospective controlled trial. Here, we aim to determine whether, in patients with a good clinical response and supratherapeutic adalimumab STLs, dose reduction based on therapeutic drug monitoring (TDM) is able to maintain the initial clinical outcome.

DETAILED DESCRIPTION:
In this study we investigate whether dose reduction of adalimumab in patients with supratherapeutic adalimumab Ctrough levels is non-inferior to standard dosing of adalimumab.

Before randomization, 3 subsequent evaluations of adalimumab Ctroughs will be executed. Patients will be included after signing informed consent and randomized if 2/3 subsequent measurements during screening show supratherapeutic Ctrough levels. Time point of randomization is considered baseline (week 0). PASI calculation will be performed by a blinded and independent physician.

In the concentration based arm, dosing frequency will be lowered to 40 mg every 3 weeks (33% reduction). In case of persistent supratherapeutic Ctroughs, a 50% dose reduction will be applied from week 12 onwards. In the standard based arm, patients will continue on standard dosing schedule of 40 mg every other week.

During each study visit PASI and IGA score will be evaluated by an independent and blinded physician and adverse events, and concomitant medications will be evaluated by a member of the study team. Ctrough is quantified at each visit; and anti-drug antibodies concentrations only if subtherapeutic concentrations are observed. Patients complete the Dermatology Life Quality Index (DLQI) and EuroQol-5D-5L instrument at each visit.

In addition, in a subset of patients in each treatment arm, additional sampling will be collected by dried blood spot sampling in order to build a PK(PD) model for adalimumab,

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be >18 years of age.
2. Participants must have a diagnosis of chronic plaque-type psoriasis for at least 6 months (with or without PsA), prior to the first administration of study intervention.
3. Participant must remain on a highly effective method of birth control during the study or during the entire treatment with adalimumab (whether with is longer)
4. Participants are considered eligible according to the following TB screening criteria:

   * Have no history of latent or active TB before screening
   * Have no signs or symptoms suggestive for active TB upon medical history and/or physical examination
   * Have had no recent close contact with a person with active TB
5. Participants must agree not to receive a live virus or live bacterial vaccination at least 3 months (or longer as indicated in the package insert of the relevant vaccine) prior to the first administration of study intervention (except for varicella and MMR vaccines), during the study, or within 3 months after the last administration of study intervention.
6. Participants must avoid prolonged sun exposure and use of tanning booths or other ultraviolet light sources during study.
7. Participants must sign an ICF indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.

Exclusion Criteria:

1. Participants who have currently a predominant nonplaque forms of psoriasis (eg. Erythrodermic, guttate, pustular)
2. Participants who are pregnant, nursing or planning a pregnancy or fathering a child while enrolled in the study or within 12 weeks after receiving the last administration of study intervention
3. Participants who have received, or are expected to receive, any live virus or bacterial vaccination (with the exception of varicella or MMR vaccines) within 3 months (or longer as indicated in the package insert of the relevant vaccine) prior to the first administration of study intervention, during the study, or within 12 weeks after the last administration of study intervention
4. Participants who have known allergies, hypersensitivity or intolerance to adalimumab or its excipients
5. Participants who have any malignancy or have a history of malignancy
6. Participants who are unable or unwilling to undergo multiple venapunctures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Clinical response | 1 year after inclusion
  The proportion of patients in each group in clinical remission (absolute PASI < 2) at year 1 after optimization
Validation of adalimumab dried blood spots | Sampling at home on days 0, 3, 5, 7, 14, 21, 28, 35, 42 and 49 after adalimumab administration
  Optimization of extraction protocol for adalimumab serum trough levels and anti-adalimumab antibody concentrations derived from dried blood spots (DBS)

SECONDARY OUTCOMES:
Relapse | 1 year after inclusion
  The proportion of patients in each group who relapse (defined as the need for dose escalation (not in the standard based dosing arm))
Serum trough levels of adalimumab within the optimal therapeutic window | 1 year after inclusion
  The proportion of patients in each group with serum trough levels (STL) of adalimumab within the optimal interval (3.5µg/ml -7 µg/ml)
Anti- drug antibodies against adalimumab | 1 year after inclusion
  The proportion of patients in each group with anti-drug antibodies (ADA) against adalimumab (ADA positivity)
Cost-effectiveness of adalimumab dose tapering | 1 year after inclusion
Quality adjusted life years | 1 year after inclusion
Identify relevant parameters for PK-PD modeling | 1 year after inclusion
  - Recording of demographic parameters during disease course monitored at baseline and at every visit (reflected by incidence, prevalence, mortality, standardized comorbidity incidence ratios and associations/risk factors).

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No